CLINICAL TRIAL: NCT04007393
Title: SMART Use of Medication for the Treatment of Adolescent Severe Obesity
Acronym: SMART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEDS-2019-26512; 1R01DK119456 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Phentermine; Topiramate

STUDY DESIGN:
Intervention Model Description: 2-staged sequential multiple assignment randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At baseline, each participant will be randomized 1:1 to either the 12-week (Arm 1) or 24-week (Arm 2) response assessment to LSMT. This randomization will be blinded to the participant, investigator, and outcomes assessor for the duration of the study; i.e. up until 48 weeks.
  The second randomization includes only those participants who are non-responders to phentermine+LSMT. Each non-responder to phentermine+LSMT will be re-randomized 1:1 to either topiramate+phentermine+LSMT or topiramate+placebo+LSMT. Participants, investigators, and outcomes assessors will be blinded to phentermine/placebo. The topiramate will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LSMT x 12 weeks (Other): Participants in this arm will start LSMT at baseline and have a weight loss response assessment at T=12 weeks: if body mass index (BMI) is down 5% at T=12 weeks, the participant will continue with LSMT for the remainder of the study (i.e. for another 36 weeks); if BMI is not down 5% at T=12 weeks, the participant will add phentermine to LSMT (phentermine+LSMT) and undergo a second weight loss response assessment after 12 weeks of phentermine+LSMT; i.e. at T=24 weeks. At T=24 weeks, if BMI is down 5% with phentermine+LSMT, the participant will continue with phentermine+LSMT for the the remainder of study (i.e. for another 24 weeks); if BMI is not down by 5% at T=24 weeks, the participant will be randomized to topiramate+phentermine+LSMT or topiramate+placebo+LSMT for the remainder of the study (i.e. for another 24 weeks).
  Interventions: Behavioral: Lifestyle Modification Therapy (LSMT); Drug: Phentermine Pill; Drug: Topiramate Pill
- LSMT x 24 weeks (Other): Participants in this arm will start LSMT at baseline and have a weight loss response assessment at T=24 weeks: if body mass index (BMI) is down 5% at T=24 weeks, the participant will continue with LSMT for the remainder of the study (i.e. for another 24 weeks); if BMI is not down 5% at T=24 weeks, the participant will add phentermine to LSMT (phentermine+LSMT) and undergo a second weight loss response assessment after 12 weeks of phentermine+LSMT; i.e. at T=36 weeks. At T=36 weeks, if BMI is down 5% with phentermine+LSMT, the participant will continue with phentermine+LSMT for the the remainder of study (i.e. for another 12 weeks); if BMI is not down by 5% at T=36 weeks, the participant will be randomized to topiramate+phentermine+LSMT or topiramate+placebo+LSMT for the remainder of the study (i.e. for another 12 weeks).
  Interventions: Behavioral: Lifestyle Modification Therapy (LSMT); Drug: Phentermine Pill; Drug: Topiramate Pill

INTERVENTIONS:
Behavioral: Lifestyle Modification Therapy (LSMT) — LSMT will consist of both in-person and by telephone sessions delivered throughout the entirety of the 48-week intervention phase. Each session will last 30-60 minutes. A trained study coordinator (a registered dietician or someone trained by our registered dietician) will delivery this therapy which consists of counseling using education, goal setting and barrier reduction. Topics covered will include calories, tracking, healthy food choices, reducing high fat, added sugar foods, setting goals and portions, changing the quality of your diet, volumetrics, purposeful activity, quick and easy meals, problem solving, food cues and eating patterns, emotional eating, accurate tracking, eating away from home, unhelpful thoughts, structured menus and the role of protein, social cues, managing stress, slips and relapse prevention, long-term physical activity and overcoming obstacles, high-risk situation and keys to success, motivation and looking to the future (long-term plans).
Drug: Phentermine Pill — Phentermine will be started only if a participant does not lose 5% of BMI after 12 or 24 weeks of LSMT depending on their random assignment. Subjects will take 15 mg of phentermine every morning for 12 weeks at which time there will be an assessment of weight loss. Subjects who achieve 5% or more BMI reduction after 12 weeks of phentermine will continue 15 mg every morning for the remainder of the study (through week 48) along with their LSMT.
Drug: Topiramate Pill — Participants who do no not achieve at least 5% BMI reduction after 12 weeks of phentermine+LSMT will be re-randomized 1:1 to either topiramate+phentermine+LSMT or topiramate+placebo+LSMT. Topiramate dosing will begin at 50 mg every morning for the first 7 days, and then increase to 100 mg every morning through week 48. At the end of week 48 the taper off will be 50 mg every morning for 7 days and then discontinue.

SUMMARY:
This study will examine the timing and sequence of using adjunct obesity pharmacotherapy for adolescents with severe obesity who do not respond to lifestyle modification therapy alone.

DETAILED DESCRIPTION:
This project is studying the best time to add weight loss medication to diet and exercise for helping adolescents who carry extra weight. All participants start with a lifestyle modification program and some participants may also receive study medication.Participants must be 12-17 years of age and carry extra weight. The program will last for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed assent form;
* Provision of signed and dated informed parental consent form from at least 1 legal parent/guardian;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* BMI >/= 1.2 times the 95th percentile or BMI >/= 35 Kg/m2, whichever is lower;
* Tanner stage >/= 2;
* Male or female, aged 12-17 at time of consenting;
* For females of reproductive potential: when sexually active, agreement to use highly effective contraception (oral contraceptive pill, intra-uterine device (IUD), or implant) during study participation;
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

* Contraindications to phentermine or topiramate use according to package inserts, including: history of glaucoma; current or recent (< 14 days) use of monoamine oxidase inhibitor; known hypersensitivity to sympathomimetic amines; current pregnancy, plans to become pregnant, or if sexually active refusal to use 2 forms of birth control; history of cardiac disease including coronary artery disease; clinically significant cardiac arrhythmias; heart failure or uncontrolled hypertension;
* Diabetes (type 1 or 2);
* Presence of cardiac pacemaker;
* Current or recent (<6 months prior to enrollment) use of weight loss medication(s);
* Current use of weight-altering medication(s) (e.g., atypical antipsychotic, metformin) unless dose has been stable for past 6 months;
* Current use of other sympathomimetic amine such as attention-deficit hyperactivity disorder (ADHD) stimulants;
* Seizure disorder (other than infantile febrile seizure);
* Previous bariatric surgery;
* Recent initiation of change in dose (< 3 months prior to enrollment) of anti-hypertensive or lipid medication(s);
* Tobacco use
* History of or current diagnosis of schizophrenia, psychosis, mania, chemical dependency;
* Unstable depression or anxiety that has required hospitalization in the past year;
* Any history of suicide attempt;
* Suicidal ideation or self-harm within 12 months prior to enrollment;
* Bicarbonate < 18 mmol/L;
* Creatinine > 1.2 mg/dL;
* History of cholelithiasis;
* History of nephrolithiasis;
* Untreated thyroid disorder;
* Hyperthyroidism;
* Breastfeeding

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Percent change in body mass index (BMI) | Baseline, 12-, 24-, 36-, and 48 weeks
  Body mass index is a measure of body fat based on height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Fox, MD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT04007393/ICF_000.pdf